CLINICAL TRIAL: NCT03285815
Title: A Phase II Randomized Trial of Hypofractionated Proton Therapy in Patients With a Localized Prostate Adenocarcinoma
Brief Title: Prostate Cancer - Localized Adenocarcinoma Proton Therapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Cancer Center, Korea (Other Government)
Responsible Party: Principal Investigator, Kwan Ho Cho, Principal Investigator, National Cancer Center, Korea
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCC 2016-0120
Record Dates: First submitted 2017-09-12; First posted 2017-09-18 (Actual); Last update posted 2017-09-18 (Actual); Status verified 2017-09

CONDITIONS: Prostate Adenocarcinoma
MeSH Terms: interventions — Proton Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Proton Therapy 60 CGE (Experimental): 60 CGE (3CGE X 20) for 4wks
  Interventions: Device: Proton Therapy
- Proton Therapy 47 CGE (Experimental): 47 CGE (4.7CGE X 10) for 2wks
  Interventions: Device: Proton Therapy

INTERVENTIONS:
Device: Proton Therapy

SUMMARY:
A Phase II Randomized Trial of Hypofractionated Proton Therapy in Patients With A Localized Prostate Adenocarcinoma

DETAILED DESCRIPTION:
For Proton therapy with prostate adenocarcinoma patients.

Arm 1: Proton therapy 3CGE x 20days = Total 60 CGE for 4 weeks.

Arm 2: Proton therapy 4.7CGE x 10days = Total 47 CGE for 2 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy proven prostate adenocarcinoma Stage: T1-T2cN0M0
* ECOG performance status:0-1
* Signed study specific informed consent prior to study entry.

Exclusion Criteria:

* Postoperative residual or recurrent tumor
* Evidence of distant metastasis previous irradiation for the tumor in the same location
* Adjuvant anti-androgenic hormonal therapy High risk group (NCCN guide line)

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 156 (Estimated)
Dates: Start 2016-05; Primary Completion 2024-05 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
BCFFS | up to 5 years from a initial follow-up
  To evaluate biochemical failure-free survival (BCFFS)

SECONDARY OUTCOMES:
Acute/late toxicity (CTCAE v4.0) | up to 5 years from a initial follow-up
  Common Terminology Criteria for Adverse Events (CTCAE) V 4.0
Disease specific survival | up to 5 years from a initial follow-up
  follow-up
EPIC (Extended Prostate Cancer Index Composite) | up to 5 years from a initial follow-up
  questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Kwanho Cho, Principal Investigator — National Cancer Center, Korea
Locations (1):
- Kwanho Cho, Ilsan, Gyenggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No